CLINICAL TRIAL: NCT01566214
Title: Representational Telehealth Nursing Intervention for Veterans With CHD
Brief Title: Vet-Harts Pilot Intervention for Veterans With Coronary Heart Disease
Acronym: VHPI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPO 09-283; 200910778 (Other: University of Iowa)
Record Dates: First submitted 2012-03-19; First posted 2012-03-29 (Estimated); Results first posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-06

CONDITIONS: Heart Disease
Keywords: coronary heart disease (CHD); myocardial infarction (MI); acute coronary syndromes (ACS)
MeSH Terms: conditions — Heart Diseases; Coronary Disease; Myocardial Infarction; Acute Coronary Syndrome | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interview (Experimental): For those subjects randomly assigned to the treatment group, information from their MIHART assessment interview and medical record review will be used to select intervention scripts optimally tailored to each subjects' unique configuration of beliefs and risk factors and they will be re-contacted by telephone at 2-weeks post-hospital discharge to deliver the Vet-HART intervention. The intervention will be administered by a trained research assistant via telephone, working from a semi-structured script tailored to each subject's representations and risk factors, the call will last about 15-30 minutes.
  Interventions: Behavioral: Motivational Interview
- Usual Care (No Intervention): For those randomly assigned to the usual care group, they will receive standard-of-care by their regular primary care provider.

INTERVENTIONS:
Behavioral: Motivational Interview — For those subjects randomly assigned to the treatment group, information from their MIHART assessment interview and medical record review will be used to select intervention scripts optimally tailored to each subjects' unique configuration of beliefs and risk factors and they will be re-contacted by telephone at 2-weeks post-hospital discharge to deliver the Vet-HART intervention. The intervention will be administered by a trained research assistant via telephone, working from a semi-structured script tailored to each subject's representations and risk factors, the call will last about 15-30 minutes.
  Arms: Motivational Interview

SUMMARY:
The purpose of this research study is to survey patients to learn about their beliefs and behaviors related to the management of heart disease and to discuss options for making healthy lifestyle changes. From the information the investigators get from patients, the investigators hope to develop better methods for taking care of patients who have heart disease.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is a significant health threat among veterans. Compared to their civilian counterparts, veterans experience greater disability, reinfarction, and mortality following myocardial infarction (MI) and other acute coronary syndromes (ACS). High rates of hypertension, diabetes, and cardiac risk behaviors (e.g., smoking) and low socioeconomic status (SES) further increase veterans' CHD-related morbidity and mortality. The proposed pilot project will establish the feasibility of a telehealth nursing intervention for veterans with CHD who are recovering from MI/ACS. The Veterans Heart Attack Representations Telehealth (Vet-HART) intervention is designed to promote adaptive conceptual change in veterans' beliefs (common sense models or representations) about CHD etiology and self-management and facilitate health behavior changes (e.g., smoking cessation, medication adherence, diet management, and increased physical activity). The long-term goal of this research program is to improve veterans' quality of life (QoL) and reduce their CHD-related morbidity/mortality. The proposed project is the requisite next step in attaining that goal.

ELIGIBILITY:
Inclusion Criteria:

* Admission to an inpatient medicine unit for MI, ACS, and coronary angiography
* Age

Exclusion Criteria:

* Altered mental status
* Language barriers
* Dementia or Cognitive Impairment
* Diagnostic Study
* Resident in long-term care facility prior to the present admission
* Planned discharge to a skilled or intermediate care facility or hospice
* Lack of access to a functioning phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2012-06-30 (Actual); Study Completion 2012-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Vander Weg, PhD MS BA, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Motivational Interview | Usual Care
Started | 6 | 6
Completed | 3 | 6
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interview | Usual Care | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.33 (11.98) | 65.67 (8.64) | 67.00 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: SF-36v Physical Function Scale
Description: Physical Functioning Subscale from the SF-36v. Possible scores range from 0 to 100, with higher scores indicating a better level of functioning.
Time Frame: Change from baseline to 3-months post hospital discharge
Population: Participants who completed the SF-36v at baseline, 1 month, and 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motivational Interview | Usual Care
Number analyzed (Participants) | 3 | 6
units on a scale | -6.67 (7.64) | 13.33 (12.52)

2. Primary Outcome: SF-36v Role Limitations Due to Physical Health Scale
Description: Role Limitations Due to Physical Health Subscale from the SF-36v. Possible scores range from 0 to 100, with higher scores indicating a better level of functioning.
Time Frame: Change from baseline to 3-months post hospital discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motivational Interview | Usual Care
Number analyzed (Participants) | 3 | 6
units on a scale | -22.92 (35.54) | 9.38 (36.39)

3. Primary Outcome: SF-36v Role Limitations Due to Emotional Problems Scale
Description: Role Limitations Due to Emotional Problems Scale from the SF-36v. Possible scores range from 0 to 100, with higher scores indicating a better level of functioning.
Time Frame: Change from baseline to 3-months post hospital discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motivational Interview | Usual Care
Number analyzed (Participants) | 3 | 6
units on a scale | -27.78 (25.46) | 5.56 (13.61)

4. Primary Outcome: SF-36v Energy-Fatigue Scale
Description: Energy-Fatigue Subscale from the SF-36v. Possible scores range from 0 to 100, with higher scores indicating a better level of functioning.
Time Frame: Change from baseline to 3-months post hospital discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motivational Interview | Usual Care
Number analyzed (Participants) | 3 | 6
units on a scale | -5.00 (42.65) | 1.67 (23.49)

5. Primary Outcome: SF-36v Emotional Well-Being Scale
Description: Emotional Well-Being Subscale from the SF-36v. Possible scores range from 0 to 100, with higher scores indicating a better level of functioning.
Time Frame: Change from baseline to 3-months post hospital discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motivational Interview | Usual Care
Number analyzed (Participants) | 3 | 6
units on a scale | -14.67 (37.86) | -2.00 (7.90)

6. Primary Outcome: SF-36v Social Functioning Scale
Description: Social Functioning Subscale from the SF-36v. Possible scores range from 0 to 100, with higher scores indicating a better level of functioning.
Time Frame: Change from baseline to 3-months post hospital discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motivational Interview | Usual Care
Number analyzed (Participants) | 3 | 6
units on a scale | -16.67 (40.18) | -10.42 (18.40)

7. Primary Outcome: SF-36v Pain Scale
Description: Pain Subscale from the SF-36v. Possible scores range from 0 to 100, with higher scores indicating a better level of functioning.
Time Frame: Change from baseline to 3-months post hospital discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motivational Interview | Usual Care
Number analyzed (Participants) | 3 | 6
units on a scale | -5.00 (13.23) | 14.17 (13.10)

8. Primary Outcome: SF-36v General Health Scale
Description: General Health Subscale from the SF-36v. Possible scores range from 0 to 100, with higher scores indicating a better level of functioning.
Time Frame: Change from baseline to 3-months post hospital discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motivational Interview | Usual Care
Number analyzed (Participants) | 3 | 6
units on a scale | -5.00 (18.03) | 4.17 (17.15)

9. Primary Outcome: Seattle Angina Questionnaire Physical Limitations Scale
Description: Physical Limitations Subscale from the Seattle Angina Questionnaire. Possible scores range from 0 to 100, with higher scores indicating a better level of functioning.
Time Frame: Change from baseline to 3-months post hospital discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motivational Interview | Usual Care
Number analyzed (Participants) | 3 | 6
units on a scale | -5.93 (8.98) | 3.33 (30.43)

10. Primary Outcome: Seattle Angina Questionnaire Angina Stability Scale
Description: Angina Stability Subscale from the Seattle Angina Questionnaire. Possible scores range from 0 to 100, with higher scores indicating a better level of functioning.
Time Frame: Change from baseline to 3-months post hospital discharge
Population: Note that because 4 participants in the Usual Care group reported that they did not experience chest pain in the prior four weeks, their responses could not be included in the analysis, as the scale measures changes in the severity of chest pain. Therefore, only 2 participants in the Usual Care group contributed to the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motivational Interview | Usual Care
Number analyzed (Participants) | 3 | 2
units on a scale | 25.00 (66.14) | -12.50 (17.68)

11. Primary Outcome: Seattle Angina Questionnaire Angina Frequency Scale
Description: Angina Frequency Subscale from the Seattle Angina Questionnaire. Possible scores range from 0 to 100, with higher scores indicating a better level of functioning.
Time Frame: Change from baseline to 3-months post hospital discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motivational Interview | Usual Care
Number analyzed (Participants) | 3 | 6
units on a scale | 20.00 (43.59) | 16.67 (22.51)

12. Primary Outcome: Seattle Angina Questionnaire Treatment Satisfaction Scale
Description: Treatment Satisfaction Subscale from the Seattle Angina Questionnaire. Possible scores range from 0 to 100, with higher scores indicating a better level of functioning.
Time Frame: Change from baseline to 3-months post hospital discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motivational Interview | Usual Care
Number analyzed (Participants) | 3 | 6
units on a scale | -3.92 (33.45) | 7.84 (10.95)

13. Primary Outcome: Seattle Angina Questionnaire Disease Perception Scale
Description: Disease Perception Subscale from the Seattle Angina Questionnaire. Possible scores range from 0 to 100, with higher scores indicating a better level of functioning.
Time Frame: Change from baseline to 3-months post hospital discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motivational Interview | Usual Care
Number analyzed (Participants) | 3 | 6
units on a scale | 13.89 (9.62) | 9.72 (17.01)

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | Motivational Interview | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No